CLINICAL TRIAL: NCT05486767
Title: Screening of Liver Fibrosis in Adults Without Known Liver Disease or With Previously Diagnosed Non-alcoholic Fatty Liver Disease
Brief Title: Screening of Liver Fibrosis in Adults Without Known Liver Disease
Acronym: SIRIUS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: F.D. Roosevelt Teaching Hospital with Policlinic Banska Bystrica (Other)
Collaborators: University Hospital Bratislava (Other); University Hospital Kosice (Unknown)
Responsible Party: Principal Investigator, Ľubomír Skladaný MD, PhD, MD, PhD, F.D. Roosevelt Teaching Hospital with Policlinic Banska Bystrica
Other Study IDs: SIRIUS
Record Dates: First submitted 2022-08-02; First posted 2022-08-04 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Liver Fibrosis
Keywords: Liver fibrosis; Screening; Non-alcoholic fatty liver disease; Alcohol associated liver disease
MeSH Terms: conditions — Liver Cirrhosis; Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool sample for microbiome analysis by 16S RNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Community cohort: SIRIUS study team will travel to pre-determined sociomes and perform transient elastography and other examinations
  Interventions: Diagnostic Test: Transient elastography
- Outpatient cohort: Patients recruited during the elective / preventive examinations at the primary-care clinics or at other outpatient-clinics will have performed Hep-calculator for FIB-4 w/wo transient elastography
  Interventions: Diagnostic Test: Transient elastography

INTERVENTIONS:
Diagnostic Test: Transient elastography — Both tests belong to the group of non-invasive tests for liver fibrosis (transient elastography belongs to the imaging-based tests and FIB-4 to the blood-based tests)
  Other Names: FIB-4 score

SUMMARY:
SIRIUS is the "serious" response to the prevalence of liver cirrhosis in Slovakia. We plan to screen adult Slovaks without acute or life-threatening comorbidity and without known liver disease (except from non-alcoholic fatty liver disease) for liver fibrosis by transient elastography (in community) or FIB-4 score (in outpatient clinics).

DETAILED DESCRIPTION:
According to the Lancet Gastroenterology and Hepatology, Slovakia ranks at the top of the prevalence of liver cirrhosis in the world. Moreover, liver diseases are the leading cause of death in the age-group of 25 - 50 years-old. SIRIUS is the response conceived by the governing board of the Slovak society of hepatology with two main aims: to screen for liver fibrosis and to spread the largely unknown information in community, and primary-care sector.

ELIGIBILITY:
Inclusion Criteria:

* adult, written informed consent

Exclusion Criteria:

* unable to provide sufficient reliable information for any reason
* withdrawal of the consent, anytime
* acute illness (e.g. febrile, drunk, on antibiotics, trauma, myocardial infarction < 2 months, operated on < 2 months, other)
* chronic disease interfering with the endpoint (malignancy < 2 years; decompensated chronic disease such as chronic heart disease with dyspnea New York heart Association NYHA 2+, Chronic obstructive pulmonary disease COPD GOLD B+, other)
* chronic liver disease other than non-alcoholic fatty liver disease without previous diagnosis of fibrosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We will approach adults of any ethnicity and gender in a stable health-status without any diseases or with a chronic extra-hepatic disease/diseases which are at the time of exam compensated and under control for more than 2 months; any medication is acceptable. Primarily, we are interested in patients without any known history of registered liver disease, but patients with steatosis without known fibrosis or cirrhosis will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-08-28 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Liver fibrosis | August, 2022 - to September 2023
  The amount of fibrous tissue in the liver according to non-invasive tests

SECONDARY OUTCOMES:
Non-alcoholic fatty liver disease | August, 2022 - September, 2023
  The amount of fat in the liver parenchyma by the non-invasive tests CAP and FLI
Alcohol associated liver disease | August, 2022 - September, 2023
  Liver disease plus AUDIT score testimonyijng to the harmful alcohol use
Body mass index | August, 2022 - September, 2023
  As calculated from height and weight (together with waist-to-hip ratio)

OTHER OUTCOMES:
Gut microbiome dysbiosis | August, 2022 - September, 2023
  Dysbiosis will be determined based on the alpha and beta diversity, followed by a the taxonomic analysis

CONTACTS AND LOCATIONS:
Overall Officials: Peter Jarčuška, Prof, Study Chair — University Hospital Košice; Martin Janičko, MD, PhD, Study Chair — University hospital Košice; Tomáš Koller, MD, PhD, Study Chair — University Hospital Bratislava
Locations (3):
- Slovakia (3):
  - F.D.Roosevelt Teaching Hospital, Banská Bystrica
  - University Hospital Bratislava, Bratislava
  - Pasteur University Hospital, Košice

IPD SHARING:
Plan to Share IPD: Yes
The whole dataset except will be shared with prof. Pere Ginés and the LiverScreen investigators
Supporting Information: Study Protocol, ICF
Time Frame: Data will be available as of December, 2023 - fo one year
Access Criteria: Consent of the SIRIUS principal investigator and chairs

REFERENCES:
- [Background] Graupera I, Thiele M, Ma AT, Serra-Burriel M, Pich J, Fabrellas N, Caballeria L, de Knegt RJ, Grgurevic I, Reichert M, Roulot D, Schattenberg JM, Pericas JM, Angeli P, Tsochatzis EA, Guha IN, Garcia-Retortillo M, Morillas RM, Hernandez R, Hoyo J, Fuentes M, Madir A, Juanola A, Soria A, Juan M, Carol M, Diaz A, Detlefsen S, Toran P, Pera G, Fournier C, Llorca A, Newsome PN, Manns M, de Koning HJ, Serra-Burriel F, Cucchietti F, Arslanow A, Korenjak M, van Kleef L, Falco JL, Kamath PS, Karlsen TH, Castera L, Lammert F, Krag A, Gines P; LiverScreen Consortium investigators. LiverScreen project: study protocol for screening for liver fibrosis in the general population in European countries. BMC Public Health. 2022 Jul 19;22(1):1385. doi: 10.1186/s12889-022-13724-6. PMID 35854275